CLINICAL TRIAL: NCT05370612
Title: Continuous Glucose Monitoring in Pregnant Patients With Type 2 Diabetes, a Mixed Methods Approach
Brief Title: AT GOAL: Adopting Technology for Glucose Optimization and Lifestyle in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-028; Protocol Version 3/18/2024 (Other: Unity Point Health - Meriter); A532860 (Other: UW Madison); 2022-0459 (Other: UW-Madison IRB)
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Type2Diabetes; Pregnancy in Diabetic
MeSH Terms: conditions — Pregnancy in Diabetics

STUDY DESIGN:
Intervention Model Description: pilot, prospective, randomized trial
Masking Description: Participant will know what arm they are randomized to, participants and physicians in Arm 2 will be blinded to CGM data collected for 10 days at 2 timepoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1: Continuous Glucose Monitor (CGM) (Experimental): CGM for duration of pregnancy.
  Interventions: Device: Dexcom G6 CGM
- Arm 2: Point of Care Glucose Testing (POCT) (Active Comparator): Point of care finger sticks for glucose monitoring.
  At two time points during the study - at time of enrollment and at 28-32 weeks gestation, CGM sensor will be placed and remain in place for 10 days. Participant and Physician will be blinded to CGM data.
  Interventions: Device: Dexcom G6 CGM; Other: Participant Finger Stick Glucose Monitoring

INTERVENTIONS:
Device: Dexcom G6 CGM — Dexcom 6 CGM, an FDA approved device. Sensors will be placed on the abdomen per package instruction to collect continuous glucose data.
  Experimental Group will wear CGM for the duration of their pregnancy.
  Control Group will have CGM data collected for 10 days at enrollment and at 28-32 weeks into their pregnancy.
Other: Participant Finger Stick Glucose Monitoring — Standard of care for individual participant
  Other Names: Glucose Monitor
  Arms: Arm 2: Point of Care Glucose Testing (POCT)

SUMMARY:
This study will assess differences in patient preferences and glucose control between continuous glucose monitoring and standard glucose checks in pregnant patients with Type 2 Diabetes. 40 participants will be on study for approximately 182 days (26 weeks).

DETAILED DESCRIPTION:
This pilot single site randomized control trial will compare the blood glucose control and participant satisfaction scores of continuous glucose monitoring vs standard glucose checks in pregnant women with a prior diagnosis of Type 2 diabetes.

The study population will consist of 40 women who are less than 20 weeks pregnant at time of enrollment who have a pre-pregnancy diagnosis of Type 2 diabetes. Participants will be randomized to one of two treatment arms.

* Arm 1: Placement of Dexcom G6 continuous glucose monitor for glucose monitoring for duration of pregnancy
* Arm 2: Continuation of standard glucose finger sticks with placement of a blinded Dexcom Pro G6 continuous glucose sensor for two ten day periods (at enrollment and again at 28-32 weeks gestation)

Participant accrual will occur over 18 months at 1 site. Participants will complete 3 study visits, all of which will be in conjunction with previously scheduled prenatal or diabetes visits: at the time of consent (less than 20 weeks gestation), 28-32 weeks gestation, and 2-6 weeks postpartum.. Surveys will be administered at each time point. At the final visit, patients will be asked for participate in a 2-5 minute directed interview as well.

* Primary Objective

  * To examine the feasibility of completing a study to assess for differences in patient preferences and glucose control between continuous glucose monitoring and standard glucose checks in pregnant patients with Type 2 Diabetes.
* Secondary Objectives

  * To estimate the effect of continuous glucose monitoring devices placed prior to 20 weeks in pregnancy in patients with Type 2 diabetes on time in range, as measured between 28-32 weeks of pregnancy.
  * To assess patient satisfaction to continuous glucose monitoring during pregnancy
  * To estimate the effect of continuous glucose monitoring on the incidence of neonatal morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age at enrollment
* Ability to consent in English
* Gestational age less than or equal to 19 weeks 6 days at enrollment
* Appropriate dating by certain LMP or ultrasound performed less than or equal to 19 weeks 6 day
* Diagnosis of Type 2 Diabetes less than or equal to 19 weeks 6 days
* Singleton gestation

Exclusion Criteria:

* Age less than 18 years of age at enrollment
* Lack of appropriate dating
* Multiple gestations
* Use of concentrated insulin at enrollment (ie U500)
* Preexisting CGM in place
* Chronic use of medications known to cause hyperglycemia, such as HIV antiretrovirals and inhaled, injectable and oral corticosteroids
* Be unwilling or unable to present to Center for Perinatal Care for visits

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-10-06 (Actual); Study Completion 2024-10-06 (Actual)

PRIMARY OUTCOMES:
Feasibility: Number of Participants Who Complete the Study within 24 month time period | up to 24 months
  Completion of the study within the 24-month timeframe, including recruitment, randomization, retention, and completion of 36 out of 40 subjects will be a measure of how feasible the intervention is.
Change in Qualitative Survey Answers to Assess Participant Thoughts and Experiences with Diabetes Management | at enrollment, 28-32 weeks gestation (up to 12 weeks on study), postpartum (up to 26 weeks on study)
  Individualized postpartum interviews and qualitative surveys administered at each time point will be used to gather information about participants thoughts and experiences in both arms of the trial about their ability to manage diabetes in pregnancy. Interviews will be analyzed for theme and content.
Percentage of Time Where Blood Glucose is between 70-140 milligrams per deciliter (mg/dL) | up to 26 weeks
  The primary endpoint is the total time within range (blood glucose level 70-140 mg/dL). All CGM data will be extracted from the Dexcom server for analysis. This measure is used to determine if time in range (TIR) is a suitable clinical endpoint for a larger trial. TIR for both arms will be determined and 95% confidence intervals around the difference in means calculated. TIR will be considered suitable if the upper 95% confidence interval for the difference in means is greater than 5 units in favor of CGM.

SECONDARY OUTCOMES:
Number of Participants with Cesarean Delivery | approximately 20 weeks on study (at time of delivery)
Change in hemoglobin A1c (percentage) from initiation to third trimester | baseline (approximately 20 weeks gestation), up to 12 weeks on study (up to 32 weeks gestation)
Percentage of time spent in hyperglycemic range | up to 26 weeks
  Hyperglycemic range is considered greater than 140 mg/dL
Percentage of time spent in hypoglycemic range | up to 26 weeks
  Hypoglycemic range is considered less than 70 mg/dL.
Rates of gestational hypertension | up to approximately 20 weeks on study
  Gestational hypertension is defined as systolic blood pressure 140 mm Hg or diastolic blood pressure 90 mg Hg on two occasions at least 4 hours apart.
Rates of preeclampsia | up to approximately 20 weeks on study
  Gestational hypertension plus either new-onset proteinuria [300 mg/24 hours, protein:creatinine 0.3 mg/dL], thrombocytopenia [platelet count<100,000/uL], elevated Aspartate transaminase or alanine transaminase [>2 upper limit of normal], renal insufficiency [serum creatinine>1.1 mg/dL or an unexplained doubling of creatinine], pulmonary edema, or cerebral or visual symptoms.
Rates of polyhydramnios | up to approximately 20 weeks on study
Incidence of neonatal hypoglycemia | up to 26 weeks
Rates of fetal macrosomia | up to 26 weeks
  Actual birthweight greater than 95 percent by Fenton growth curve for newborns
Rates of NICU Admission | up to 26 weeks
Rates of spontaneous preterm delivery | up to approximately 17 weeks on study (less than 37 weeks gestation)
  Preterm delivery is considered less than 37 weeks.
Satisfaction and Quality of Life Survey Scores (5-point likert scale) | at enrollment, 28-32 weeks gestation (10 to 14 weeks on study), 2-4 weeks postpartum (up to 26 weeks on study)
  A custom survey for Satisfaction and Quality of Life will be administered and answers will be compared between groups. Survey questions include answers on a 5-point likert scale, 7-point likert scale, and participant count data. Survey questions scored on a 5-point likert scale are reported here where higher scores indicated increased satisfaction and quality of life.
Satisfaction and Quality of Life Survey Scores (7-point likert scale) | at enrollment, 28-32 weeks gestation (10 to 14 weeks on study), 2-4 weeks postpartum (up to 26 weeks on study)
  A custom survey for Satisfaction and Quality of Life will be administered and answers will be compared between groups. Survey questions include answers on a 5-point likert scale, 7-point likert scale, and participant count data. Survey questions scored on a 7-point likert scale are reported here where higher scores indicated increased satisfaction and quality of life.
Satisfaction and Quality of Life Survey Scores (Participant Counts) | at enrollment, 28-32 weeks gestation (10 to 14 weeks on study), 2-4 weeks postpartum (up to 26 weeks on study)
  A custom survey for Satisfaction and Quality of Life will be administered and answers will be compared between groups. Survey questions include answers on a 5-point likert scale, 7-point likert scale, and participant count data. Survey questions scored as participant counts are reported here.
Qualitative Outcome: Semi-Structured Interviews to Explore How Glucose Monitoring Affects Participants Thoughts and Feelings | 2-4 weeks postpartum (up to 26 weeks on study)
  The interviews will be recorded and transcribed by the Survey Center and analyzed for theme and content by two reviewers for validity.
Qualitative Outcome: Interviews to understand Participant Sense of Control around Glucose Monitoring | 2-4 weeks postpartum (up to 26 weeks on study)
  Explore if traditional management versus continuous glucose management has higher feelings of control over diabetes management. The interviews will be recorded and transcribed by the Survey Center and analyzed for theme and content by two reviewers for validity.

CONTACTS AND LOCATIONS:
Overall Officials: Jacquelyn H Adams, MD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No